CLINICAL TRIAL: NCT01131442
Title: Immunological Change and the Single Nucleotide Polymorphism (SNP) in Children With Irritable Bowel Syndrome (IBS)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Chang Gung Memorial Hospital, Chang Gung Memorial Hospital
Other Study IDs: CMRPG270371
Record Dates: First submitted 2010-05-25; First posted 2010-05-27 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2010-05

CONDITIONS: Irritable Bowel Syndrome; Children
Keywords: immune
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- The patient group
- healthy control group

SUMMARY:
Currently, the pathophysiology of Irritable bowel syndrome( IBS) remains unclear . The purpose of this study is want to investigate the immunological changes in the children with IBS.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is a highly prevalent functional gastrointestinal disorder.Many children suffered from this disease and had impact on their daily life. However, the underlying pathophysiologic mechanisms remain to be elucidate. Dysregulation of the gut immune system is considered an important pathophysiology. We want to investigate the immunological changes in the IBS children.

ELIGIBILITY:
Inclusion Criteria:

* (5-18y/o) with IBS,
* All patients had chronic or relapsing symptoms of IBS consistent with the ROME II criteria

Exclusion Criteria:

* A history of psychologic disorders, probiotics, anti-inflammatory, analgesic, or immunosuppressive medication (nonsteroidal anti-inflammatory drugs, steroids) within the past 3 months were excluded

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: out patient clinics in the hospital
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2008-11

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memeorial Hospital, Keelung, Taiwan

REFERENCES:
- [Derived] Hua MC, Chao HC, Yao TC, Lai MW, Huang JL; PATCH Study Group. Investigation of interleukin-10 promoter polymorphisms and interleukin-10 levels in children with irritable bowel syndrome. Gut Liver. 2013 Jul;7(4):430-6. doi: 10.5009/gnl.2013.7.4.430. Epub 2013 Jun 11. PMID 23898383
- [Derived] Hua MC, Lai MW, Kuo ML, Yao TC, Huang JL, Chen SM. Decreased interleukin-10 secretion by peripheral blood mononuclear cells in children with irritable bowel syndrome. J Pediatr Gastroenterol Nutr. 2011 Apr;52(4):376-81. doi: 10.1097/MPG.0b013e3181fd9816. PMID 21407110